CLINICAL TRIAL: NCT00957970
Title: Periprosthetic Bone Mineral Changes Around Stemless and Stemmed Cementless Femoral Components
Brief Title: Bone Mineral Changes Around Stemless and Stemmed Cementless Femoral Components
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Young-Hoo, Kim M.D., Ewha Womans University Mokdong Hospital Joint Replacement Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009-7-17
Record Dates: First submitted 2009-07-21; First posted 2009-08-13 (Estimated); Last update posted 2009-08-13 (Estimated); Status verified 2009-08

CONDITIONS: Osteoarthritis of Hip
Keywords: Stress shielding; Bone mineral density; stemless femoral component
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stemless femoral component (Active Comparator): Stemless PROXIMA femoral component
  Interventions: Device: Stemless femoral component
- Stemmed femoral component (Active Comparator): IPS, proximal anatomical fit stemmed femoral component
  Interventions: Device: IPS, Depuy cementless femoral stem

INTERVENTIONS:
Device: Stemless femoral component — Total hip femoral component anatomically designed for a proximal fit without a stem
  Other Names: PROXIMA, DePuy stem,
  Arms: Stemless femoral component
Device: IPS, Depuy cementless femoral stem — Anatomical proximal fitted cementless stemmed femoral component
  Other Names: IPS, Depuy anatomical proximal fit stemmed femoral component
  Arms: Stemmed femoral component

SUMMARY:
The purpose of this study is to determine if there is a difference in stress shielding and bone resorption of the proximal femur in two anatomical stem total hip designs.

DETAILED DESCRIPTION:
Stress shielding related bone resorption in the proximal femur after total hip arthroplasty continues to be a problem. The purpose of this prospective, randomized study was to evaluate which of the two anatomical stem designs achieved a more physiological load transfer by assessing bone mineral changes in the proximal femur after stem implantation.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis of hip joint requiring total hip arthroplasty

Exclusion Criteria:

* Neurologic disorders affecting motor function of lower extremity
* foot and ankle disorders limiting ambulation of the patient
* Patients with bone metabolic disorders other than osteoporosis which prevents normal bone metabolism
* Multi-systemic inflammatory arthritis which debilitates patients other than hip joint.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-07; Primary Completion 2007-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Bone mineral density of surrounding proximal femur according to Gruen zones | At least 2years after surgery

SECONDARY OUTCOMES:
Harris hip score | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Young-Hoo Kim, MD, Study Director — Korean Joint replacement Center
Locations (1):
- Ewha Womans University Mokdong Hospital, Seoul, South Korea

REFERENCES:
- [Background] Gulow J, Scholz R, Freiherr von Salis-Soglio G. [Short-stemmed endoprostheses in total hip arthroplasty]. Orthopade. 2007 Apr;36(4):353-9. doi: 10.1007/s00132-007-1071-x. German. PMID 17377765
- [Background] Albanese CV, Santori FS, Pavan L, Learmonth ID, Passariello R. Periprosthetic DXA after total hip arthroplasty with short vs. ultra-short custom-made femoral stems: 37 patients followed for 3 years. Acta Orthop. 2009 Jun;80(3):291-7. doi: 10.3109/17453670903074467. PMID 19562565
- [Background] Renkawitz T, Santori FS, Grifka J, Valverde C, Morlock MM, Learmonth ID. A new short uncemented, proximally fixed anatomic femoral implant with a prominent lateral flare: design rationals and study design of an international clinical trial. BMC Musculoskelet Disord. 2008 Nov 4;9:147. doi: 10.1186/1471-2474-9-147. PMID 18983669
- [Background] Kim YH. Cementless total hip arthroplasty with a close proximal fit and short tapered distal stem (third-generation) prosthesis. J Arthroplasty. 2002 Oct;17(7):841-50. doi: 10.1054/arth.2002.33555. PMID 12375241